CLINICAL TRIAL: NCT01136460
Title: Genetic Testing in Primary Congenital Glaucoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, Professor, Carmel Medical Center
Other Study IDs: CMC052005CTIL
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Congenital Glaucoma
Keywords: Primary congenital glaucoma; neonatal; Genotype correlation; Phenotype correlation
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primary congenital glaucoma: Primary congenital glaucoma patients and their immediate relatives

SUMMARY:
Primary congenital glaucoma patients and their immediate relatives will undergo complete ophthalmic examination and an interview with a geneticist. A blood sample will be drown from all participants for DNA analysis.

The CYP1B1 gene coding sequences will be screened for all individuals. If no mutation or only one heterozygous mutation will be found in the CYP1B1 gene, screening for MYOC gene mutations will be performed.

DETAILED DESCRIPTION:
Primary congenital glaucoma (PCG) is usually present in the neonatal or

infantile period and is accompanied by corneal opacity and edema, buphthalmos, increased intraocular pressure, optic nerve cupping, and at times, ensuing severe visual impairment. The incidence of the disease varies significantly in different geographic regions and is more frequently found in certain ethnic groups, especially where consanguinity is prevalent. The incidence in Western countries has been reported to range from 1:5000 and 1:10000 births, and in populations where consanguinity is prevalent, such as among Slovakian Gypsies and Saudi Arabians, the incidence ranges from 1:1250 and 1:2500 births, respectively. PCG is believed to be an autosomal-recessive transmitted disease with incomplete penetrance. Three different loci have been mapped for it, i.e., GLC3A on chromosome 2p21, GLC3B on 1p36.2 and GLC3C on 14q24.3. The major gene that currently has been identified to be associated with PCG is the CYP1B1 gene at locus GLC3A, which encodes a member of the cytochrome P450. The frequency of mutations in the CYP1B1 gene in PCG patients varies in different geographic locations and ethnic groups. For example, mutations in the CYP1B1 gene are found in 33% of patients in Japan and Indonesia, while among Saudi Arabian and Slovakian Gypsy patients, the incidence rises to 94% and 100%, respectively. Mutations in myocilin (MYOC) have also been associated with PCG.

Determining the presence of CYP1B1 mutations in PCG patients will improve our ability to counsel parents regarding cause, inheritance and the risk of it in future offspring.

The aim of the present study is to characterize the phenotype and determine the role of CYP1B1 and MYOC mutations in PCG in Israeli populations

ELIGIBILITY:
Inclusion Criteria:

* Primary congenital glaucoma pediatric patients
* Glaucoma that was diagnosed within the first 12 months of their life
* Primary congenital glaucoma pediatric patients's parents

Exclusion Criteria:

* any other ocular or systemic diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary congenital glaucoma patients and their immediate relatives
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2006-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Mutations in the CYP1B1 gene | one year
  Mutations in the CYP1B1 gene were detected in 12 of 26 (46%) families with PCG (5 Muslim Arab, 5 Druze, 2 Jewish). Jewish families had compound heterozygous mutations, i.e. an Ashkenazi family had mutations in the CYP1B1 gene (Arg368His and R48G, A119S and L432V haplotypes), and an Ashkenazi-Sephardic family had a mutation on the CYP1B1 gene (1908delA, Sephardic) with a second missense mutation on the MYOC gene (R76K, Ashkenazi). Muslim Arabs and Druze tended to have a more severe phenotype than did the Jews.

CONTACTS AND LOCATIONS:
Overall Officials: Orna Geyer, Professor, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Geyer O, Wolf A, Levinger E, Harari-Shacham A, Walton DS, Shochat C, Korem S, Bercovich D. Genotype/phenotype correlation in primary congenital glaucoma patients from different ethnic groups of the Israeli population. Am J Ophthalmol. 2011 Feb;151(2):263-71.e1. doi: 10.1016/j.ajo.2010.08.038. Epub 2010 Dec 18. PMID 21168818